CLINICAL TRIAL: NCT04665648
Title: Impact of Intravenous Administration of Nicorandil As Adjuncts to Reperfusion Treatment for Acute ST Segment Elevation Myocardial Infarction: a Multi-center Randomized Controlled Trial
Brief Title: Clinical Efficacy and SAfety of Intravenous Infusion of Nicorandil During Primary Percutaneous Coronary Intervention
Acronym: CLEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ge Junbo, Director, Dept. of Cardiology, Zhongshan Hospital, Fudan University, Shanghai, China, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-CLEAN
Record Dates: First submitted 2020-12-02; First posted 2020-12-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: ST Elevation Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Patients who received intravenous nicorandil before and after reperfusion with primary percutaneous coronary intervention
  Interventions: Drug: Nicorandil
- Placebo arm (Placebo Comparator): Patients who received intravenous placebo before and after reperfusion with primary primary percutaneous coronary intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicorandil — 6 mg nicorandil iv. just before coronary intervention, 6mg/h ivgtt. up to 48h after coronary intervention
  Other Names: intraveous nicorandil
  Arms: Treatment arm
Drug: Placebo — placebo iv. just before coronary intervention, ivgtt. up to 48h after coronary intervention
  Other Names: intraveous palcebo
  Arms: Placebo arm

SUMMARY:
The investigators evaluate the efficacy and safety of intravenous administration of nicorandil as adjuncts to reperfusion treatment in acute ST-segment elevation acute myocardial infarction (STEMI) patients undergoing primary percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years;
* acute ST-segment elevation myocardial infarction within 12 hours of symptom onset;

Exclusion Criteria:

* systolic blood pressure<100mmHg;
* cardiac shock;
* aortic dissection;
* history of myocardial infarction or percutaneous coronary intervention or coronary artery bypass grafting (<6 month);
* history of the treatment of nicorandil (<6 month);
* history of intravenous nitrates before percutaneous coronary intervention;
* contraindicated or intolerable to nicorandil;
* pregnant or lactation period;
* patients with an estimated survival time of less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 12 month after primary PCI
  cardiac death, myocardial reinfarction, target vessel revascularization, unplanned hospitalization for heart failure

SECONDARY OUTCOMES:
Rate of slow re-flow/no-reflow | 3 minutes after primary PCI
  final coronary flow in the culprit artery
Rate fo complete ST-segment resolution | 2 hours after primary PCI
  ST-segment resolution >50% in ECG
Cardiac death | 12 months after primary PCI
  Cardiac death
Myocardial reinfarction | 12 months after primary PCI
  Myocardial reinfarction
Target vessel revascularization | 12 months after primary PCI
  Target vessel revascularization
Unplanned hospitalization for heart failure | 12 months after primary PCI
  Unplanned hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of the summary data
Access Criteria: IPD collected in this study generated or analyzed during the study are available from the corresponding author by request.

REFERENCES:
- [Background] Kitakaze M, Asakura M, Kim J, Shintani Y, Asanuma H, Hamasaki T, Seguchi O, Myoishi M, Minamino T, Ohara T, Nagai Y, Nanto S, Watanabe K, Fukuzawa S, Hirayama A, Nakamura N, Kimura K, Fujii K, Ishihara M, Saito Y, Tomoike H, Kitamura S; J-WIND investigators. Human atrial natriuretic peptide and nicorandil as adjuncts to reperfusion treatment for acute myocardial infarction (J-WIND): two randomised trials. Lancet. 2007 Oct 27;370(9597):1483-93. doi: 10.1016/S0140-6736(07)61634-1. PMID 17964349
- [Background] Kawai Y, Hisamatsu K, Matsubara H, Dan K, Akagi S, Miyaji K, Munemasa M, Fujimoto Y, Kusano KF, Ohe T. Intravenous administration of nicorandil immediately before percutaneous coronary intervention can prevent slow coronary flow phenomenon. Eur Heart J. 2009 Apr;30(7):765-72. doi: 10.1093/eurheartj/ehp077. Epub 2009 Mar 10. PMID 19276198
- [Background] Wu M, Huang Z, Xie H, Zhou Z. Nicorandil in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention: a systematic review and meta-analysis. PLoS One. 2013 Oct 22;8(10):e78231. doi: 10.1371/journal.pone.0078231. eCollection 2013. PMID 24167609
- [Derived] Huang D, Wu H, Zhou J, Zhong X, Gao W, Ma Y, Qian J, Ge J. Intravenous nicorandil during primary percutaneous coronary intervention in patients with ST-Elevation myocardial infarction: Rationale and design of the Clinical Efficacy and Safety of Intravenous Nicorandil (CLEAN) trial. Am Heart J. 2022 Feb;244:86-93. doi: 10.1016/j.ahj.2021.11.005. Epub 2021 Nov 14. PMID 34785173